CLINICAL TRIAL: NCT06370351
Title: A Phase I/II, Open-ended, Adaptative, Open Label Dose Escalation and Expansion Clinical Trial to Evaluate the Efficacy and Safety of Unilateral Intracochlear Injection of SENS-501 Using an Injection System in Children with Severe to Profound Hearing Loss Due to Otoferlin Gene Mutations
Brief Title: A Phase I/II Clinical Trial with SENS-501 in Children Suffering from Severe to Profound Hearing Loss Due to Otoferlin (OTOF) Mutations
Acronym: AUDIOGENE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SENS-501-101; 2023-504466-28-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: OTOF Gene Mutation; DFNB9; Congenital Deafness; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases; Deafness; Hearing Loss, Sensorineural
Keywords: OTOF Gene Mutation; Hearing impairment; Deafness; otoferlin; AUDIOGENE; Hearing Loss; DFNB9; Hearing disorder; Cochlear implant; SENS-501; Congenital Hearing loss; Gene therapy
MeSH Terms: conditions — Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases; Deafness; Hearing Loss, Sensorineural; Hearing Loss; Deafness, Autosomal Recessive 9

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation - Low dose group (Experimental): Intracochlear administration of a Low dose of SENS-501 in one ear, with a dedicated administration system
  Interventions: Combination Product: SENS-501 administration
- Dose escalation - High dose group (Experimental): Intracochlear administration of a High dose of SENS-501 in one ear, with a dedicated administration system
  Interventions: Combination Product: SENS-501 administration
- Dose expansion group (Experimental): Intracochlear administration of SENS-501 in one ear, with a dedicated administration system, at the dose recommended following the Dose escalation phase
  Interventions: Combination Product: SENS-501 administration

INTERVENTIONS:
Combination Product: SENS-501 administration — Administration of SENS-501 with a dedicated administration system

SUMMARY:
This study intends to assess safety, tolerability, and efficacy of SENS-501 in children between the ages of 6-31 months with pre-lingual hearing loss due to a mutation in the Otoferlin gene.

DETAILED DESCRIPTION:
It is a multicenter, adaptive open-label, non-randomized, dose-escalation, and expansion study to assess safety, tolerability, and efficacy following intracochlear administration of SENS-501.

ELIGIBILITY:
Inclusion Criteria:

* Children (male or female) ≥ 6 to ≤ 31 months at the time of inclusion
* Severe to profound hearing loss assessed by auditory brainstem response (ABR)
* Biallelic mutation in the Otoferlin gene
* Presence of Otoacoustic emissions (OAEs)
* Documented normal cochlea and internal auditory canals
* Patients with intact vestibular function

Exclusion Criteria:

* History of chronic, acute, or major disease, or unspecified reasons, that in the opinion of the Investigator, makes the participant unsuitable for participation in the study or constitutes an unacceptable risk.
* Have been dosed in a previous gene therapy clinical trial
* Patients with a prior or current cochlear implant
* Any contraindication to the surgery determined by the surgeon or anesthesia determined by the anesthesiologist, or designee, or history of therapy known as ototoxic (e.g., cisplatin, high dose and long treatment with aminoglycosides, etc.) for an extended period (more than 2 weeks).
* Participation in any other interventional clinical trial
* Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the participant or would preclude the participant from successful completion of the study or might interfere with the evaluation of study treatment
* Anticipated noncompliance with the protocol requirements

Ages: 6 Months to 31 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SENS-501 | 5 years
  Number of study-related adverse events (AEs) and serious adverse events (SAEs).
Efficacy of SENS-501 assessed by ABR | 5 years
  Improvement of hearing threshold measured by auditory brainstem response (ABR)

SECONDARY OUTCOMES:
Safety and tolerability of SENS-501 | 5 years
  Number of study-related adverse events (AEs) and serious adverse events (SAEs).
Efficacy of SENS-501 assessed by ABR | 5 years
  Improvement of hearing threshold measured by auditory brainstem response (ABR)
Efficacy of SENS-501 assessed by PTA | 5 years
  Improvement of hearing threshold measured by Pure-tone audiometry (PTA)
Clinical performance of the administration system | 1 day
  Administration success ; Users' feedback questionnaire on the administration and use of the devices
Safety of the administration system | 5 years
  Adverse device effects and Device deficiencies, Procedure complications
Usability of the administration system | 1 day
  Usability questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Natalie LOUNDON, Pr, Study Chair — Hopital Necker Enfants Malades
Locations (2):
- Childrens Hospital Westmead, Westmead, Australia
- Hopital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No